CLINICAL TRIAL: NCT04763681
Title: Expanding a Randomized Controlled Trial of a Couple Internet-Delivered PTSD Intervention to Reach Military Members, Veterans, and First Responders With COVID-19-Related Trauma Exposure
Brief Title: Couple HOPES (Helping Overcome PTSD and Enhance Satisfaction)
Acronym: HOPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Skye Fitzpatrick, Assistant Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-475; 173098 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); CIHR-IRSC:0525007697 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); W7714-207266 (Other Grant/Funding Number: National Defence Security Orders and Directives)
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Self-help; Internet-delivered intervention; Couple satisfaction; COVID-19; Coronavirus
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Participating couples are randomized to either immediately receive the Internet-delivered Couple HOPES intervention or to a delayed intervention group, where they receive access to Couple HOPES 8 weeks later.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Couple HOPES (Experimental): Immediately assigned to receive seven modules of an Internet-delivered self-help intervention with paraprofessional coaching for PTSD completed at the participant's own pace within 8 weeks.
  Interventions: Behavioral: Couple HOPES Guided, Internet-Delivered, Self-Help Intervention
- Delayed Intervention (No Intervention): Participants will not receive Couple HOPES for the first 8 weeks, and complete assessments at the beginning, middle, and end of this period. After this 8-week delay, participants will then receive seven modules of an Internet-delivered self-help intervention with paraprofessional coaching for PTSD completed at the participant's own pace within 8 weeks.

INTERVENTIONS:
Behavioral: Couple HOPES Guided, Internet-Delivered, Self-Help Intervention — Couple HOPES is a guided self-help intervention for individuals with PTSD and their partners based on Cognitive-Behavioral Conjoint Therapy for PTSD (Monson & Fredman, 2012). This intervention consists of text and video-based content across seven intervention modules and phone and online-based coaching sessions with a paraprofessional. Participants are able to complete these modules in their own home or private location of their choosing. The primary outcomes are PTSD symptoms, relationship satisfaction, and the mental health and wellbeing of partners of those with PTSD.
  Arms: Immediate Couple HOPES

SUMMARY:
Posttraumatic Stress Disorder (PTSD) will be a severe problem in Canada in the wake of COVID-19, especially for Military Members, Veterans, First Responders, and Healthcare Workers (MVFH). However, gold standard face-to-face PTSD treatments do not meet current MVFH needs, which requires virtual interventions and minimal healthcare resources. Recognizing the need for a virtual, low-resource PTSD intervention for MVFH with PTSD and their loved ones, the investigators developed Couple HOPES (Helping Overcome PTSD and Enhance Satisfaction). Couple HOPES is a secure, online self-help intervention for those with PTSD and their partners (www.couplehopes.com). However, MVFH are now particularly likely to be exposed to traumas related to COVID-19. It is essential to identify if Couple HOPES is safe and helpful for couples involving MVFH with COVID-19-related PTSD specifically. This project will therefore test the efficacy of Couple HOPES compared to a delayed waitlist control in 70 couples wherein one member is a MVFH with COVID-19-related PTSD. The investigators will examine if Couple HOPES is helpful in improving PTSD symptoms and relationship satisfaction for such couples, and if it is more or less helpful to this end for these couples compared to those with other forms of trauma exposure. 70 couples including a MVFH with COVID-19-related PTSD, will be randomly assigned to receive Couple HOPES or to a waitlist. PTSD symptoms and relationship satisfaction will be measured ~weekly during the intervention and one month after it. Related problems (e.g., depression, anxiety, healthcare use) will be measured before, in the middle of, after, and one month after, the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individual who is a Canadian military member, veteran, first responder or healthcare worker with clinically significant levels of PTSD symptoms related to COVID-19
* Individual who is an American healthcare worker with clinically significant levels of PTSD symptoms related to COVID-19
* Must be willing to be audio-recorded for coaching sessions
* Intimate partner willing to participant and complete intervention modules together
* Access to high speed internet

Exclusion Criteria:

* Elevated suicide risk
* Severe physical aggression between partners in the past year
* Clinically significant PTSD symptoms in both members of the dyad

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5) with change measured as mean change from baseline | Baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, and 3 months after the intervention
  Scores on the PCL-5 range from 0 to 80, with 80 being the most severe PTSD symptoms.
Couple Satisfaction Index (CSI-4) with change measured as mean change from baseline | Baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, and 3 months after the intervention
  Score on the CSI-4 range from 0 to 21, with 21 being the most satisfied.

SECONDARY OUTCOMES:
Mean change from baseline on Ineffective Arguing Inventory | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Score range from 0 to 40, with 40 representing highly ineffective arguing.
Significant Others' Responses to Trauma Scale with change measured as mean change from baseline | Baseline, week 3, week 8, 3 month post-treatment follow-up
  Scores range from 0 to 76, with 76 representing high partner accommodation.

OTHER OUTCOMES:
Mean change from baseline on depression as measured by the Patient Health Questionnaire | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 27, with 27 being the most depressed.
Mean change from baseline on alcohol use as measured by the Alcohol Use Disorders Identification Test: Self-Report Version | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 40, with a higher score signifying an alcohol use disorder.
Mean change from baseline in drug use based on the Drug Abuse Screen Test | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 10, with 10 being a severe level of problems related to drug abuse.
Generalized Anxiety Disorder symptoms with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 21, with 21 representing the highest level of anxiety.
State-Trait Anger Expression Inventory with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 0 to 40, with 40 representing higher levels of anger.
Mean change from baseline in perceived health measured with one item "How satisfied are you with your health" | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
  Scores range from 1 to 5, with 5 being the most satisfied.
Trauma-Related Guilt Inventory with change measured as mean change from baseline | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Mean change from baseline in work functioning measured with one item "Please rate your ability to function at work. If you do not work outside the home, please rate your ability to complete household tasks." | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Mean change from baseline in quality of life measured with one item "How would you rate your quality of life." | Baseline, week 3, week 8, after 3 modules are completed or 3 weeks into treatment, after 7 modules are completed or 8 weeks into treatment, 3 month post-treatment follow-up
Participant ratings of intervention satisfaction as indicated by the Client Satisfaction Questionnaire | After 7 modules are completed or 8 weeks into treatment
Feasibility as measured by number of treatment sessions attended and rate of participant dropout | Once a week during treatment (for up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Skye Fitzpatrick, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monson, C. M., & Fredman, S. J. (2012). Cognitive-behavioral conjoint therapy for PTSD: Harnessing the healing power of relationships. New York, NY: Guilford.
- [Derived] Fitzpatrick S, Crenshaw AO, Valela R, Samonas C, Earle EA, Goss S, Hernandez KM, Bushe J, Varma S, Proctor D, Wagner AC, Goenka K, Luxor O, Collins A, Morland L, Shields N, Roth M, Doss BD, Schumm J, Monson CM. A randomized controlled trial testing couple HOPES: An online, self-help couples' intervention for posttraumatic stress disorder. J Consult Clin Psychol. 2025 Aug;93(8):580-594. doi: 10.1037/ccp0000965. PMID 40811121